CLINICAL TRIAL: NCT07325682
Title: Personalized, Scientifically Based Technologies in the Diagnosis and Treatment of SARS-CoV-2 as a Possible Cervical Cancer Risk Factor
Brief Title: Diagnostic Evaluation of Viral Persistence in Cervical Cancer
Acronym: PETCVOCC
Status: Enrolling by invitation | Phase: Not Applicable | Type: Interventional
Sponsor: Oncology Center,Ministry Of Heath,Uzbekistan (Other)
Responsible Party: Principal Investigator, Naylya Djumaeva, Principal Investigator, Oncology Center,Ministry Of Heath,Uzbekistan
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: CC-DIAG-001
Record Dates: First submitted 2025-12-09; First posted 2026-01-08 (Actual); Last update posted 2026-01-08 (Actual); Status verified 2025-12

CONDITIONS: Cervical Cancer
Keywords: medicament testing; viral antigen persistance; Human Papillomavirus
MeSH Terms: conditions — Uterine Cervical Neoplasms

STUDY DESIGN:
Masking Description: Diagnostic evaluation of viral persistence using EAV-based measurement of viral activity in cervical cancer patients.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Diagnostic Group (Experimental): Non-invasive diagnostic method assessing bioelectrical response patterns associated with viral markers in patients with cervical cancer.
  Interventions: Diagnostic Test: Electroacupuncture

INTERVENTIONS:
Diagnostic Test: Electroacupuncture — Non-invasive electrodiagnostic assessment using electroacupuncture measurements to evaluate bioelectrical response patterns associated with viral markers in patients with cervical cancer.

SUMMARY:
This study aims to evaluate the diagnostic value of an electroacupuncture-based method for detecting viral persistence (human papillomavirus and SARS-CoV-2) in patients with cervical cancer. The study investigates whether persistent viral signatures can be identified through measurable electrodiagnostic responses at acupuncture points associated with organ systems affected by chronic viral infection. The goal is to assess the feasibility, reproducibility, and potential clinical relevance of this diagnostic approach in oncology patients.

DETAILED DESCRIPTION:
This study investigates the diagnostic potential of an electroacupuncture-based measurement method to detect viral persistence in patients with cervical cancer. Increasing evidence indicates that oncologic processes may be influenced by chronic viral activity, including persistent human papillomavirus (HPV) infection and, in some cases, secondary viral signatures such as SARS-CoV-2. Although HPV is the primary etiologic agent in cervical cancer, clinical observations suggest that long-term viral presence may contribute to variations in disease behavior, immune dysfunction, and treatment response.

The diagnostic method used in this study is based on measurement of electrical parameters at standardized acupuncture points. These points are functionally connected to organ systems involved in chronic viral disease. Changes in their electrical characteristics may reflect physiological responses associated with viral persistence. The technique has been previously developed and refined in clinical practice and has demonstrated reproducibility in identifying characteristic response patterns in patients with viral and post-viral conditions.

This study aims to evaluate whether measurable electrodiagnostic responses correlate with persistent viral signatures in cervical cancer patients. All participants undergo standardized diagnostic measurements performed under controlled conditions. The study does not involve therapeutic intervention, drug administration, or device implantation. Only diagnostic data are collected.

The primary objective is to assess whether this method can reliably identify patterns consistent with viral persistence. Secondary objectives include evaluating repeatability of measurements, describing characteristic profiles in this patient population, and assessing feasibility of integrating this diagnostic approach into clinical oncology settings.

This research is expected to contribute to a better understanding of viral involvement in cancer microenvironments and to support the development of non-invasive diagnostic tools for evaluating viral activity in oncologic patients.

ELIGIBILITY:
Inclusion Criteria:

* Histologically confirmed cervical cancer (FIGO stage IIIA-IVA)
* Age ≥21 years
* ECOG performance status adequate for diagnostic procedures
* Adequate organ function
* Ability to provide informed consent

Exclusion Criteria:

* Poor renal function (elevated creatinine)
* Significant liver dysfunction (elevated bilirubin or liver enzymes)
* Severe cardiovascular or pulmonary disease
* Pregnancy or breastfeeding
* Severe mental illness or inability to provide informed consent
* Known non-compliance or substance abuse

Ages: 21 Years to 70 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2025-04-30 (Actual); Primary Completion 2026-06-30 (Estimated); Study Completion 2030-12-30 (Estimated)

PRIMARY OUTCOMES:
Number of Participants With Bioelectrical Patterns Consistent With Viral Antigen Persistence | At enrollment (single diagnostic session)
  Diagnostic assessment to identify bioelectrical response patterns associated with viral antigen persistence in cervical cancer patients using a non-invasive bioelectrical testing approach.

CONTACTS AND LOCATIONS:
Locations (1):
- City Branch of the National Oncology and Radiology Center, Tashkent, Uzbekistan

IPD SHARING:
Plan to Share IPD: No
Individual participant data (IPD) will not be shared because the study involves a small diagnostic cohort and contains sensitive clinical information that cannot be anonymized to a level ensuring full participant privacy. The data will be used only for internal scientific analysis within the approved protocol.